CLINICAL TRIAL: NCT05410041
Title: Safety and Efficacy of Anti-CD19 CAR-Engineered NK Cells for Relapsed/Refractory B-cell Malignancies: a Multi-center, Open-label, Single-arm Clinical Study
Brief Title: Anti-CD19 CAR-Engineered NK Cells in the Treatment of Relapsed/Refractory B-cell Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Boren Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRYY-IIT-LCYJ-2022-003
Record Dates: First submitted 2022-05-26; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Acute Lymphocytic Leukemia; Chronic Lymphocytic Leukemia; Non Hodgkin Lymphoma
Keywords: CAR-NK; CD19 positive; B-cell malignancy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-NK-CD19 Cells (Experimental): After preconditioning with chemotherapy, CAR-NK-CD19 Cells will be evaluated.
  Interventions: Biological: CAR-NK-CD19 Cells

INTERVENTIONS:
Biological: CAR-NK-CD19 Cells — CAR-NK-CD19 Cells, 1-3×10^7 /KG, treatment follows a lymphodepletion. Drug: Fludarabine Recommendation: 25-30 mg/kg (D-5~D-3), determined by tumor burden at baseline. Drug: Cyclophosphamide Recommendation: 250-300 mg/kg (D-5~D-3), determined by tumor burden at baseline.

SUMMARY:
This study is a single arm, open and multi center exploratory clinical study to observe the safety and effectiveness of CAR NK-CD19 in participants with recurrent or refractory CD19 positive B-cell malignant tumors, and preliminarily evaluate the expansion of this product in vivo and the objective remission rate after administration.

DETAILED DESCRIPTION:
The study will enroll 9-21 participants diagnosed with recurrent or refractory CD19 positive B-cell malignant tumors, including acute B-lymphocyte leukemia, B-cell non-Hodgkin's lymphoma and chronic B-lymphocyte leukemia. There will be three preset dose groups in this clinical trial, which are 1.0×10^7、2.0×10^7 and 3.0×10^7 CAR positive NK cells / kg (body weight), SRC will discuss and decide the next infusion plan. Participants will be enrolled from low dose group to high dose group, each dose will enroll at least 3 cases. Dose escalation will be decided by the SRC (Safety Review Committee) separately by diseases. There will be expanded cases in the aim dose group, which will at most to 6 cases. The protocol will be performed into screening period (-30~-10 days), prophase of lymophodepletion (-10~-5 days), Lymophodepletion (-5~-3 days), pre-infusion evaluation (-2~-1 days), infusion (day 0), and follow-up period (1-720 days). According to the administration strategy, we will start from single administration. Only after the SRC's decision based on safety and PK data, we could explore further on multiple administrations or combo therapy strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, regardless of gender;
2. Eastern Cooperative Oncology Group score 0-2;
3. Participants with CD19 positive B-cell malignancies, including acute lymphocytic leukemia (all), chronic lymphocytic leukemia (CLL) and non-Hodgkin lymphoma (NHL);
4. Failure or recurrence of at least 2-line treatment (including immunotherapy, targeted therapy and stem cell transplantation);
5. Measurable lesions with an expected survival of more than 3 months;
6. The functions of liver, kidney, heart and lung meet the following requirements:

   * creatinine clearance rate ≥ 60ml / min ;
   * ALT (alanine transaminase, ALT) / AST (aspartate aminotransferase, AST) ≤ 2.5 times the upper normal limit;
   * total bilirubin ≤ 1.5 times the upper limit of normal value, except for participants with Gilbert syndrome, the total bilirubin must be < / = 3.0 mg / dl;
   * left ventricular ejection fraction ≥ 50%, no clinically significant ECG results;
   * blood oxygen saturation > 92% in non oxygen absorption state;
7. The subjects agreed to use reliable contraceptive methods for contraception within 1 year from the signing of informed consent to reinfusion. Including but not limited to: abstinence, male vasectomy, implantable progesterone contraceptives that can inhibit ovulation; Intrauterine device; Hormone releasing intrauterine device; Sexual partner sterilization; Copper IUD, correct use of proven compound hormone contraceptives that can inhibit ovulation; Progesterone contraceptives that inhibit ovulation. At the same time, the subjects should promise not to donate eggs (oocytes, oocytes) / sperm for assisted reproduction within 1 year after reinfusion;
8. Voluntarily participate in clinical trials and sign informed consent.

Exclusion Criteria:

1. Known allergic reaction, hypersensitivity, intolerance or contraindication to CAR NK-CD19 or any component of drugs that may be used in the study (including fludarabine, cyclophosphamide and tozumab), or subjects who have had severe allergic reaction in the past;
2. Participants with gastrointestinal lymph nodes and / or central nervous system involvement who were judged by the researchers to be at risk by CAR NK-CD19 treatment (except those who were judged by the researchers to be more likely to benefit than risk);
3. Those who have graft-versus-host response and need to use immunosuppressants; or suffering from autoimmune diseases;
4. Before screening, the researchers judged that corticosteroids needed to receive a long-term therapeutic dose during the study period;
5. Received the following anti-tumor treatment within the specified time before screening:

   i. Have received small molecule targeted therapy within 4 weeks or 5 half lives (whichever is longer); ii. Have received macromolecular drug treatment within 4 weeks or 2 half lives (whichever is longer); iii. Have received cytotoxic treatment or modern traditional Chinese medicine preparation with antitumor effect within 2 weeks;
6. Those who have been vaccinated with live vaccine or attenuated vaccine within 4 weeks before screening; Note: it is allowed to receive inactivated virus vaccine for seasonal influenza; However, it is not allowed to receive live attenuated influenza vaccine for intranasal use;
7. History of epilepsy or other central nervous system diseases;
8. Other active malignant tumors in the two years before screening (except for the following cases: tumors targeted in this study, surgically removed non-melanoma skin cancer, cured cervical carcinoma in situ, local prostate cancer, low-stage bladder cancer, breast ductal carcinoma in situ, or no recurrence and no treatment of malignant tumors in the two years before randomization);
9. Within 14 days before enrollment, there were active or uncontrollable infections requiring systemic treatment;
10. Active hepatitis B participants; Hepatitis C virus (HCV) antibody positive; Human immunodeficiency virus (HIV) antibody positive; Syphilis antibody positive in primary screening;

    a) Participants with inactive / asymptomatic carrier, chronic or active HBV infection can be included if they meet the following conditions: HBV DNA < 500 IU / ml (or 2500 copies / ml) at the time of screening.
11. The toxicity (including peripheral neuropathy) caused by previous treatment has not fully recovered or stabilized to grade 1 (nci-ctcae V5.0) (except those that the researcher judges will not affect the patient's safe treatment, such as hair loss);
12. Heart disease: there is heart failure (NYHA classification ≥ class II, Appendix 2) and serious heart disease determined by the researcher; Myocardial infarction occurred ≤ 6 months before screening; Unstable angina pectoris, severe arrhythmia judged by the researcher or coronary artery bypass grafting (CABG) occurred ≤ 3 months before screening;
13. Poor control of hypertension (systolic blood pressure > 160 mmHg and / or diastolic blood pressure > 100 mmHg) or accompanied by hypertensive crisis or hypertensive encephalopathy;
14. Participants who had undergone major surgery or plasma separation other than diagnosis or biopsy within 4 weeks before screening, or were expected to undergo major surgery during the study; Note: participants who plan to perform surgery under local anesthesia can participate in the study. Kyphoplasty or laminoplasty is not considered a major operation;
15. Those who are receiving thrombolytic, anticoagulant or antiplatelet therapy;
16. The subjects judged by the researcher are difficult to complete all visits or operations required by the study protocol, or the compliance of participating in the study is insufficient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Safety of CAR NK-CD19 Cell | Up to 3 months after cell infusion
  Safety of CAR NK-CD19 will be assessed by incidence and severity of AEs and SAEs.
The overall response rate (ORR) | Up to 3 months after cell infusion
  Objective response rate (ORR) according to NCCN, Complete response(CR),CR with incomplete blood count recovery(CRi).

SECONDARY OUTCOMES:
Concentration of PK CAR positive NK cells in peripheral blood | Up to 3 months after cell infusion
  PK CAR positive NK cells in peripheral blood, PK CAR transgene levels in peripheral blood
Pharmacodynamic data in peripheral blood | Up to 3 months after cell infusion
  The amount and duration of antibody to CAR NK-CD19 cells in peripheral blood.

OTHER OUTCOMES:
Duration of remission (DOR) after infusion | From 28 to 180 days after infusion
  refers to the time from the first assessment of CR or PR to the first assessment of disease progression or death from any cause
Progression-free survival (PFS) after infusion | From 28 to 180 days after infusion
  refers to the time from cell infusion to the first assessment of tumor progression or recurrence or death from any cause
Overall survival (OS) after infusion | From 6 to 24 months after infusion
  refers to the time from cell infusion to death due to any cause. For subjects who have dropped out before death, the dates of their last visit would be counted as their time of death; if the subject receives other new treatments, the time of death will be calculated based on the start date of the new treatment; if the study ends, the time of death will be calculated based on the end date

CONTACTS AND LOCATIONS:
Overall Officials: Kai Hu, MD/PhD, Principal Investigator — Beijing Boren Hospital
Locations (1):
- Beijing Boren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No